CLINICAL TRIAL: NCT01779713
Title: Discovery of the Risk Factors Associated to the Development of Vasospasm Following a Sub-arachnoid Aneurismal Hemorrhage Via Genomic Studies Including Genetic and Transcriptomic
Brief Title: Transcriptomic Signature of Vasospasm Consecutive to Sub-arachnoid Aneurismal Hemorrhage
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C10-15; 2012-A00935-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2013-01-10; First posted 2013-01-30 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2022-02

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Vasospasm
Keywords: Aneurysmal subarachnoid hemorrhage; Vasospasm; Transcriptomic; Case-Control Study
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vasospastic patients: Any patient send to the neuro-anesthesia intensive care unit in the 48 hours following an aneurismal sub-arachnoid hemorrhage and treated in the 96 first hours (embolization or surgery) and developing a vasospasm during the first 12 days after the bleeding; aged more than 18; of Caucasian origin; affiliated to a social care service; having (or one of is related if he is comatose) given its informed consent
  Interventions: Genetic: Case-control transcriptomic study
- Control patients: Any patient send to the neuro-anesthesia intensive care unit in the 48 hours following an aneurismal sub-arachnoid hemorrhage and treated in the 96 first hours (embolization or surgery) not developing a vasospasm during the first 12 days after the bleeding; aged more than 18; of Caucasian origin; affiliated to a social care service; having (or one of is related if he is comatose) given its informed consent
  Interventions: Genetic: Case-control transcriptomic study

INTERVENTIONS:
Genetic: Case-control transcriptomic study — No intervention

SUMMARY:
Rational: The main danger with intracranial aneurism is its rupture conjugated with subarachnoid hemorrhage (SAH) occurrence. SAH is a severe pathology leading not only to neurological but also extra cerebral disorders. The major cause of morbidity and mortality when developing a SAH is the secondary development of a delayed cerebral ischemia consecutive to a prolonged vasospasm of cerebral arteries. The understanding of the pathophysiological mechanisms of SAH complication, such as vasospasm which is the more frequent, is essential.

Vasospasm is defined as a reversible shrinking of an artery lumen diameter in the subarachnoid space, beginning generally between 4 and 12 days after the hemorrhage. Such a vasospasm could have a huge clinical impact leading to delayed neurological ischemic deficiency in 17 to 40 % of cases. Up to day, mechanisms involved in vasospasm occurrence are not well described.

Disposing of well-established genetics and transcriptomics databases along with cerebral ischemia and inflammation is essential to unravel the mechanisms leading to vasospasm occurrence on SAH patients. It will enable researchers to better comprehend SAH pathology and elaborate an efficient and individualized therapeutic strategy to SAH acute phase in order to reduce the risk of vasospasm occurrence.

Aims: 1) Constitute DNA and RNA Biobank via blood proofing oh SAH patients 2) Constitute a database grouping clinical and biological data 3) Look for genetic and transcriptomic early markers via genomic approaches 4) Correlate these different markers with vasospasm occurrence and clinical evolution of the patients

Study: Patients inclusion will be done following their admission (D1) in the " unité de réanimation neurochirurgicale" of Pitié-Salpètrière Hospital. After obtaining of the informed consent, blood proofing will be realized daily during 12 days: one daily 2.5ml tube for the transcriptomic study and a single 10ml EDTA tube for genetic analyses. Clinical and biological follow-up will be performed as usual.

200 patients will be initially included during 2 to 3 years for the transcriptomic study of which 1/3 will develop vasospastic complication. The transcriptomic study will thus be performed by comparing patients developing or not developing this complication

Expected Results: Unravel vasospasm early genetic markers.

ELIGIBILITY:
Inclusion Criteria:

* Patient entering the neurosurgical unit in the 48 hours following an aneurismal sub-arachnoid hemorrhage and treated in the 96 first hours (embolization or surgery)
* Aged more than 18
* Caucasian origin
* Affiliated to a social care service
* Having (or one of is related if he is comatose) given its informed consent

Exclusion Criteria:

* Subjects which do not have a social care protection
* Subjects (or one of is related if he is comatose) refusing to sign the consent
* Subjects being under a protective juridical system for adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caucasian subjects, aged more than 18, suffering of sub-arachnoid hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Evidence of clinically definite vasospasm | Between intensive care unit admission and day twelve
  Any cases will be reviewed by an expert committee to establish vasospasm diagnosis
  Diagnosis criteria:
  * Cerebral angiography,
  * Trans-cranial Doppler of the MCA at 120 cm/s or two days of changing in the mean speed of the MCA at trans-cranial Doppler superior to 50 cm/s.
  * Development of new clinical symptoms for conscious patients

SECONDARY OUTCOMES:
Rankin Score | 6 months and 1 year after ICU discharge
Glasgow outcome score (GOS) | 6 months and 1 year after ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Garnier, Lecturer, Study Director — INSERM and University Pierre and Marie Curie; Louis Puybasset, MD PhD, Study Chair — Pierre and Marie Curie University
Locations (1):
- Neuro-anesthesia intensive care unit, Pitié-Salpétrière hospital, Paris, France

REFERENCES:
- [Result] Pulcrano-Nicolas AS, Proust C, Clarencon F, Jacquens A, Perret C, Roux M, Shotar E, Thibord F, Puybasset L, Garnier S, Degos V, Tregouet DA. Whole-Blood miRNA Sequencing Profiling for Vasospasm in Patients With Aneurysmal Subarachnoid Hemorrhage. Stroke. 2018 Sep;49(9):2220-2223. doi: 10.1161/STROKEAHA.118.021101. PMID 30354977
- [Result] Pulcrano-Nicolas AS, Jacquens A, Proust C, Clarencon F, Perret C, Shotar E, Puybasset L, Le Goff W, Degos V, Tregouet DA, Garnier S. Whole blood levels of S1PR4 mRNA associated with cerebral vasospasm after aneurysmal subarachnoid hemorrhage. J Neurosurg. 2019 Nov 29;133(6):1837-1841. doi: 10.3171/2019.9.JNS191305. Print 2020 Dec 1. PMID 31783362